CLINICAL TRIAL: NCT03901664
Title: Lymphocyte Sub-populations and Auto Immune Diseases : What Type of Profile ? (SPLIT)
Brief Title: Lymphocyte Sub-populations and Auto Immune Diseases
Acronym: SPLIT
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SPLIT ( 29BRC17.0243)
Record Dates: First submitted 2018-12-04; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2018-09

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine if artificial intelligence allow to detect lymphocyte subpopulations specific of diseases (such as primary Sjogren' syndrome and systemic lupus erythematosus) among patients with suspicion of autoimmune diseases.

DETAILED DESCRIPTION:
The goal of this study is to determine if artificial intelligence allow to detect lymphocyte subpopulations specific of diseases (such as primary Sjogren' syndrome and systemic lupus erythematosus) among patients with suspicion of autoimmune diseases.

All patients who had an evaluation of their lymphocyte subpopulations between january 2010 and december 2016 will be included in a retrospective analysis.

ELIGIBILITY:
Inclusion Criteria:

* autoimmune or infectious disease

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: autoimmune diseases (lupus and Sjogren's) or chonic infection (Whipple's disease)
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of autoimmune disease | an average of 1 year
  Diagnosis (systemic lupus erythematosus, primary Sjopgren's ....) according to current ACR/EULAR criteria

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France